CLINICAL TRIAL: NCT05320484
Title: The Effect Of Clinical Pilates Exercises On Posture In The Adult Patients With Shoulder-Neck Posture Problem: A Single-blind Randomized Controlled Trial
Brief Title: Clinical Pilates Exercises On Posture In Patients With Shoulder-Neck Posture Problem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meltem Uzun (Other)
Responsible Party: Sponsor-Investigator, Meltem Uzun, Director, Sanko University
Organization: Sanko University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MeltemU
Record Dates: First submitted 2022-03-22; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Posture; Exercise
Keywords: Posture; Head and Shoulder; Pilates Based Exercises
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clinical pilates exercises (Experimental): clinical pilates exercises applied to 1st group,for 3 days / week for 6 weeks.
  Interventions: Other: Clinical Pilates Exercises
- classical posture exercises (Other): classical postural exercises applied to 2 nd group,for 3 days / week for 6 weeks.
  Interventions: Other: Classic Posture exercise

INTERVENTIONS:
Other: Clinical Pilates Exercises — clinical pilates exercises methods applied to the 1st group, classical posture exercises methods to the 2nd group for 3 days / week for 6 weeks.
  Arms: clinical pilates exercises
Other: Classic Posture exercise — clinical pilates exercises methods applied to the 1st group, classical posture exercises methods to the 2nd group for 3 days / week for 6 weeks.
  Arms: classical posture exercises

SUMMARY:
This study was designed to investigate the effect of clinic pilates exercise in adult patients whith shoulder- neck posture problem. 51 patients with forward head posture(FHP) and rounded shoulder posture(RSP) were included in this study and they were randomly divided into two groups as clinical pilates (group 1, n=26) and classical posture exercises (group 2, n=25). Patients' demographics were recorded. Deep neck fleksor muscle(DNFM) endurance was evaluated by pressure biofeedback unit (PBU). Head, neck and shoulder posture were evaluated with wall- tragus, wall-acromion, tragus-acromion and chin-sternal notch distance. Flexibility for shoulder region was evaluated with back scratch test. The patients were evaluated both before the study and 6 weeks later.

DETAILED DESCRIPTION:
Fifty-one individuals aged between 20-55 years whose FHP and RSP problems were determined by lateral posture analysis were included in the study. However, a total of 12 individuals, 6 from each of the 2 groups, were excluded from the study because they could not complete the treatment sessions. The study was completed with 39 participants.Individuals aged between 20-60 years, whose FHP and RSP problems were determined by lateral posture analysis, were included in the study. Those with severe pain in the neck and shoulder girdle, scoliosis and neurological problems and those who had undergone any surgery in the relevant regions were not included in the study. The individuals included in the study were randomized by lot and divided into 2 groups. Group 1 was given clinical pilates exercises, and Group 2 was given a program consisting of classical posture exercises. The exercise programs of both groups were performed by the same physiotherapist, and pre- and post-exercise evaluations were made by a different physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* FHP and RSP problems were determined by lateral posture analysis

Exclusion Criteria:

* skoliosis

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-06-18 (Actual); Study Completion 2017-07-18 (Actual)

PRIMARY OUTCOMES:
Distance Measurements | 6 week
  The right-left tragus-wall distance, right-left tragus-acromion distance, right-left wall-acromion distance, and chin-sternal notch distance were measured with the help of a tape measure.
The DNFM endurance | 6 week
  The DNFM endurance of the cases was measured using a pressurized biofeedback unit (PBU
Shoulder Region Flexibility | 6 week
  Back Scratch Test

CONTACTS AND LOCATIONS:
Overall Officials: Meltem uzun, Study Director — Sanko University
Locations (1):
- SANKO University, Gaziantep, Please Select, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No